CLINICAL TRIAL: NCT01424267
Title: Zenith® LP AAA Endovascular Graft Post-Market Registry
Brief Title: Zenith® LP Abdominal Aortic Aneurysm (AAA) Post-Market Registry
Status: Terminated | Type: Observational
Why Stopped: The registry was discontinued due to significant resources required.
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-006
Record Dates: First submitted 2011-08-23; First posted 2011-08-26 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Abdominal Aortic Aneurysm; Aorto-iliac Aneurysm
Keywords: low profile; endovascular graft; endovascular procedure; aortic aneurysm, abdominal aortic aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1
  Interventions: Device: Zenith® Low Profile AAA Endovascular Graft

INTERVENTIONS:
Device: Zenith® Low Profile AAA Endovascular Graft — Treatment of an abdominal aortic or aorto-iliac aneurysm with the CE-marked Zenith(R) Low Profile AAA Endovascular Graft.

SUMMARY:
A registry to collect additional prospective intra-operative and follow-up information on physician use of the CE-marked Zenith® Low Profile Abdominal Aortic Aneurysm (AAA) Endovascular Graft under routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Patient is implanted with Zenith® Low Profile AAA Endovascular Graft

Exclusion Criteria:

* Patients for whom this device would not normally be considered standard of care.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients implanted with a CE-Marked Zenith® Low Profile AAA Endovascular Graft
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2010-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
graft patency and aneurysm exclusion | during (day 1) and after implantation through 12 months

CONTACTS AND LOCATIONS:
Locations (15):
- AKH (General Hospital Vienna), Vienna, Austria
- Germany (3):
  - UHZ Hamburg GmbH (Eppendorf University Hospital), Hamburg
  - Klinikum rechts der Isar (RDI Munich), Munich
  - Klinikum Nürnberg Süd, Nuremberg
- Royal Victoria Hospital, Belfast, Ireland
- Italy (2):
  - Nuovo Ospendale Civile Sant' Agostino Estense di Baggiovara, Modena
  - Azoemda ospedaliera San Camillo Forlanini, Rome
- Netherlands (2):
  - Catharina Ziekenhuis, Eindhoven
  - Maastricht University Medical Center, Maastricht
- St. Olav University Hospital, Trondheim, Norway
- United Kingdom (5):
  - Guy's and St. Thomas' Hospital, London
  - St. Mary's Hospital, London
  - Manchester Royal Informary, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Royal Gwent Hospital, Wales